CLINICAL TRIAL: NCT04320563
Title: Efficacy and Safety of Rexon Eye in Asian Dry Eye
Brief Title: Rexon-Eye in Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R1624/21/2019; 2019/2446 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye
Keywords: Rexon-eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the participants and Investigators were masked. Only the study staff we helped with the Rexon-eye treatment was unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full power treatment 4 (Active Comparator): These group of participants will receive the full power treatment 4
  Interventions: Procedure: Rexon-eye
- Comparative Power 1 (Placebo Comparator): These group of participants will receive the comparative power 1 treatment
  Interventions: Procedure: Rexon-eye

INTERVENTIONS:
Procedure: Rexon-eye — This treatment involved the technology known as quantum molecular resonance (QMR) which has emerged as a new treatment for all types of dry eyes.

SUMMARY:
Resono Ophthalmic has developed Rexo-Eye in 2014, a QMR-based patented instrument which is hypothesised to stimulate physiological cellular regeneration and reactivate the tear system by stimulating and reactivating the lacrimal system, induce mild hyperthermia and massage effects which reactivate the tear and lipid secretion, targeting all arms of pathogenic mechanisms of dry eye disease. By improving cell migration and cell health, eye surface epithelial problems in dry eyes which are hard to reverse could hopefully be improved. It has been marked since 2016 as a medical device for the treatment of ocular surface disorders and patented in Italy and Europe, with other international patents pending. In this study, we aim to assess the efficacy and safety of Rexon-Eye in dry eye patients.

DETAILED DESCRIPTION:
Dry eye disease, or ocular surface disease (OSD)as defined by the International Dry Eye Workshop (2007)1, is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance and tear film instability with potential damage to the ocular surface.1

There is an armantaranium of therapies different types of dry eyes such as lubricating eyedrops, moisture retention chamber, intense pulsed light which are not curative and require repetitive application. Recently, Quantum molecular resonance (QMR) has emerged as a new treatment for all types of dry eyes. This technology involves transpalpebral non-invasive high frequency microcurrent electrical stimulation of cells which stimulate natural regeneration of cells. With the application of low-power high-frequency oscillating electrical currents in the range of 4 to 64 megahertz, it works via the resonance effect by maximising delivery of energy to biological tissues by oscillating electrical fields without increasing temperature and eliciting biological responses.2, 3 A previous in-vitro study had evaluated the biophysical effects these high frequency electrical fields on cells in culture, which showed that it invoked a series of cellular massage of contractions and relaxations' which trigger cellular metabolism and stimulate tissues.

Resono Ophthalmic has developed Rexo-Eye in 2014, a QMR-based patented instrument which is hypothesised to stimulate physiological cellular regeneration and reactivate the tear system by stimulating and reactivating the lacrimal system, induce mild hyperthermia and massage effects which reactivate the tear and lipid secretion, targeting all arms of pathogenic mechanisms of dry eye disease. By improving cell migration and cell health, eye surface epithelial problems in dry eyes which are hard to reverse could hopefully be improved. It has been marked since 2016 as a medical device for the treatment of ocular surface disorders and patented in Italy and Europe, with other international patents pending. Therapy takes place in the form of special mask electrodes applied to the patient's periorbital area worn for 20 minutes per session.

Earlier studies have shown evidence to improve subjective and objective symptoms of dry eye disease as well as to successfully reduce the number of tear substitute eye drops over a 2 month treatment period with Rexon-Eye. However, these studies are mainly small scale and conducted in Western populations. There have been no other studies conducted in Asian populations on the efficacy and safety of the Rexon-Eye device in targeting dry eye disease. Thus our study aims to evaluate these two aims through this study, while determining patient satisfaction and acceptability of the technology and furthermore, exploring changes in the composite of tears before and after the Rexon-Eye device.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old and above;
2. Diagnosed with moderate dry eyes based on grade 3 and worse corneal fluorescein staining in the central interpalpebral region
3. Are on other eye drops (including artificial tears, topical ciclosporin, steroids), blephagel or lid warming solely for dry eyes, with no recent change in the last 1 month;
4. Willing to perform all eye examinations in this study;
5. Clear of exclusion criteria

Exclusion Criteria:

1. Pregnant women
2. Patients carrying active implantable device (e.g., pacemakers and hearing aids)
3. Oncologic patients under treatment
4. Patient who underwent ocular surgery in the last month
5. Patients who are vegan or exclude egg in their diet
6. Patient who is on antibiotic or glaucoma eye drops
7. Patient who had ocular infection within 6 months
8. Any other specified reason as determined by clinical investigator

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
SPEED Questionnaire to access the dry eye symptoms | 3 months
  To assess the improvement of dry eye symptoms by SPEED questionnaire

SECONDARY OUTCOMES:
Acceptance of treatment (Rexon-eye) | 3 months
  Participants will be asked to answer some questions on the satisfaction and acceptability of Rexon-eye treatment

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No